CLINICAL TRIAL: NCT00536068
Title: Platelet Inhibition by Aspirin, Acetaminophen and NSAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Graubünden (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KGWR0206
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-09-28 (Estimated); Status verified 2007-09

CONDITIONS: Hemostasis
Keywords: platelet; aggregation; aspirin
MeSH Terms: interventions — Aspirin; Acetaminophen; Diclofenac; Naproxen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1, 2, 3, 4 (Experimental): 1. acetylsalicylic acid 100 mg/po,acetaminophen 3x1g/po
  2. acetylsalicylic acid 100 mg/po,diclofenac 3x50mg/po
  3. acetylsalicylic acid 100 mg/po,naproxen 3x250mg/po
  4. acetylsalicylic acid 100 mg/po,placebo 3x1/po
  Interventions: Drug: Acetylsalicylic acid, acetaminophen, diclofenac, naproxen, placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid, acetaminophen, diclofenac, naproxen, placebo — 1. Acetylsalicylic acid 100mg/po and acetaminophen 3x1g/po for 4 days
  2. Acetylsalicylic acid 100mg/po and diclofenac 3x50mg/po for 4 days
  3. Acetylsalicylic acid 100mg/po and naproxen 3x250mg/po for 4 days
  4. Acetylsalicylic acid 100mg/po and placebo 3x1/po for 4 days

SUMMARY:
Nonsteroidal antiinflammatory drugs such as diclofenac or naproxen may interfere with the inhibition of platelet aggregation by aspirin, because they all interact with the platelet cyclooxygenase.This may be of great clinical importance because of an increased cardiovascular event rate (myocardial infarction, stroke). The present randomized, controlled study analyses in vitro platelet aggregation under a combined treatment of healthy volunteers with aspirin and either acetaminophen, diclofenac, naproxen, or placebo.

DETAILED DESCRIPTION:
An in vivo study on healthy volunteers with combinations of well established drugs

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Administration of drugs affecting platelets
* History of bleeding
* Gastrointestinal disorders
* Hypersensitivity to aspirin and/or NSAID
* Pregnancy and breast feeding

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
platelet aggregation | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Walter H Reinhart, MD Professor, Principal Investigator — Department of Internal Medicine, Kantonsspital Graubunden CH7000 Chur Switzerland
Locations (1):
- Kantonsspital Graubünden, Department of Internal Medicine, Chur, Switzerland